CLINICAL TRIAL: NCT00448435
Title: A Study to Compare GW815SF HFA MDI With Concomitant Treatment With Salmeterol Xinafoate DPI Plus Fluticasone Propionate DPI and to Assess Long-term Safety of GW815SF HFA MDI
Brief Title: Clinical Assessment Of GW815SF HFA MDI In Pediatric Patients With Bronchial Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 110099
Record Dates: First submitted 2007-03-14; First posted 2007-03-16 (Estimated); Results first posted 2009-08-11 (Estimated); Last update posted 2010-06-08 (Estimated); Status verified 2010-06

CONDITIONS: Bronchial Asthma
Keywords: Salmeterol; Fluticasone propionate; Salmeterol/Fluticasone propionate combination; Pediatric bronchial asthma
MeSH Terms: conditions — Asthma | interventions — Fluticasone-Salmeterol Drug Combination

ARMS (3):
- SLM+FP First (Active Comparator): SLM(salmeterol) 25mcg + FP(fluticasone propionate) 50mcg twice daily in first intervention period and SFC(salmeterol/fluticasone propionate) 25/50mcg twice daily in second intervention period and (after washout period).
  Interventions: Drug: GW815SF HFA MDI; Drug: salmeterol and fluticasone propionate
- SFC First (Active Comparator): SFC (Salmeterol/Fluticasone propionate combination) 25/50mcg twice daily in first intervention period and SLM (Salmeterol) 25mcg + FP (Fluticasone Propionate) 50mcg twice daily in second intervention period (after washout period).
  Interventions: Drug: GW815SF HFA MDI; Drug: salmeterol and fluticasone propionate
- SFC (Experimental): SFC (salmeterol/fluticasone propionate combination) 25/50mcg twice daily in Extension period (after cross-over period).
  Interventions: Drug: GW815SF HFA MDI

INTERVENTIONS:
Drug: GW815SF HFA MDI — salmeterol and fluticasone propionate combination
  Other Names: salmeterol/fluticasone propionate combination
Drug: salmeterol and fluticasone propionate — salmeterol + fluticasone propionate
  Arms: SFC First; SLM+FP First

SUMMARY:
To evaluate the efficacy and safety of GW815SF HFA MDI 25/50µg 1 inhalation bid in comparison with concomitant treatment with salmeterol xinafoate DPI 25µg 1 inhalation bid plus fluticasone propionate DPI 50µg 1 inhalation bid in paediatric patients with asthma.

To evaluate the safety of long-term treatment of GW815SF HFA MDI 25/50µg 1 inhalation bid in paediatric patients with asthma.

ELIGIBILITY:
Inclusion criteria:

* Inclusion Criteria for Entry in Run-in Period

A pediatric patient already diagnosed as having bronchial asthma who meets all of the following criteria is eligible for the study:

* Male or female patients aged ≥5 and ≤14 years. Enrolment of a female patient of childbearing potential is allowed only if she is tested negative in the pregnancy testing at the start of Treatment Period 1 and if she agrees to undergo pregnancy testing at the protocol-specified timings and to take contraceptive measures without fail.
* Written informed consent must be obtained from a legally acceptable representative of the subject. Consent of the subject him/herself should also be obtained, wherever possible, after giving an explanation in an as easy to understand as possible manner.
* An outpatient who has been treated with ICS (FP 100μg/day or equivalent) for at least 4 weeks prior to Visit 1.
* Able to use a peak flow meter in a correct manner in the investigator's/subinvestigator's judgment.
* Able to use MDI and DPI in a correct manner (with the assistance of his/her caregiver as necessary) in the investigator's/subinvestigator's judgment.

Inclusion Criteria for Entry in Treatment Period 1 A subject will be randomized to one of the two treatment groups only if he/she has completed the run-in period and meets all the following criteria.

1. Has a mean of morning PEF measurements in the last 7 days of the run-in period (excluding the first day of Treatment Period 1) ≤90% of his/her best PEF measurement .
2. Was able to perform entry in the asthma diary and PEF measurements in a correct manner in the investigator's/subinvestigator's judgment.
3. Able to use MDI and DPI in a correct manner (with the assistance of his/her caregiver as necessary) in the investigator's/subinvestigator's judgment.

Exclusion criteria:

* Exclusion Criteria for Entry in Run-in Period

A patient who applies any of the following criteria is not eligible for the study:

* Admitted to the hospital due to asthma exacerbation within 8 weeks prior to Visit 1.
* Used systemic steroid within 4 weeks prior to Visit 1.
* Received antibacterials or antivirals for treatment of upper or lower respiratory tract infection within 2 weeks prior to Visit 1.
* Has a safety problem in participation in the study because of a serious, uncontrolled systemic disease including nervous system disorder.
* Has or is suspected to have deep-seated mycosis or infection to which no effective antibacterial agent is available.
* Has or is suspected to have hypersensitivity to the investigational product, rescue medication or any ingredients of them.
* Is pregnant or lactating, may be pregnant, or plans for pregnancy during the study period.
* Has received the last dose in another clinical study within 2 months prior to this study.
* Is not eligible for the study in the investigator's/subinvestigator's judgment.

Exclusion Criteria for Entry in Treatment Period 1

Enrolment of a subject completing the run-in period into Treatment Period 1 will not be allowed if any of the following applies:

1. Admitted to the hospital due to asthma exacerbation during the run-in period.
2. Had upper or lower respiratory tract infection during the 2 weeks just before Visit 2.
3. Used prohibited drugs during the 2 weeks just before Visit 2.
4. Is not eligible for the study in the investigator's/subinvestigator's judgment.

Exclusion Criteria for Entry in Treatment Period 2

Enrolment of a subject completing the washout period into Treatment Period 2 will not be allowed if any of the following applies:

1. Admitted to the hospital due to asthma exacerbation during the washout period.
2. Had upper or lower respiratory tract infection during the 2 weeks just before Visit 4.
3. Used prohibited drugs during the 2 weeks just before Visit 4.
4. Is not eligible for entry in Treatment Period 2 in the investigator's/subinvestigator's judgment.

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2007-04; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- Japan (4):
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Saitama
  - GSK Investigational Site, Tokyo

RESULTS

PARTICIPANT FLOW:
Groups:
- SFC 50/100 Mcg/Day First: GW815SF (SFC; Salmeterol/Fluticasone propionate combination) HFA (Hydro Fluoro Alkane) MDI (Metered Dose Inhaler) 25/50 mcg twice daily in first intervention period and SLM (Salmeterol) DPI (Dry Powder Inhaler) 25 mcg + FP (Fluticasone Propionate) DPI 50 mcg twice daily in second intervention period (after washout period).
- SLM 50 Mcg + FP 100 Mcg/Day First: SLM (Salmeterol) DPI (Dry Powder Inhaler) 25 mcg + FP (Fluticasone Propionate) DPI 50 mcg twice daily in first intervention period and GW815SF (SFC; Salmeterol/Fluticasone Propionate combination) HFA (Hydro Fluoro Alkane) MDI (Metered Dose Inhaler) 25/50 mcg twice daily in second intervention period (after washout period).
Period: Treatment Period I - 4 Weeks
Arm/Group | SFC 50/100 Mcg/Day First | SLM 50 Mcg + FP 100 Mcg/Day First
Started | 26 | 25
Completed | 26 | 25
Not Completed | 0 | 0
Period: Washout Period - 2 Weeks
Arm/Group | SFC 50/100 Mcg/Day First | SLM 50 Mcg + FP 100 Mcg/Day First
Started | 26 | 25
Completed | 25 | 25
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Treatment Period II - 4 Weeks
Arm/Group | SFC 50/100 Mcg/Day First | SLM 50 Mcg + FP 100 Mcg/Day First
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0
Period: Extension Period - 20 Weeks
Arm/Group | SFC 50/100 Mcg/Day First | SLM 50 Mcg + FP 100 Mcg/Day First
Started | 50 | 0
Completed | 50 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study Population: Randomized Population
Arm/Group | Overall Study Population
Number analyzed (Participants) | 51
Age Continuous [Mean (Standard Deviation); unit: Years] | 8.3 (2.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 34
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian-Japanese Heritage | 51
Region of Enrollment [Number; unit: participants]
  Japan | 51

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Mean Change From Baseline in Morning PEF (Peak Expiratory Flow) During the 4-week Treatment Periods
Description: Mean change from baseline = value at each assessment period (mean of the values obtained at each assessment period [Weeks 1-4/Weeks 7-10]) minus baseline value. Baseline: Mean of the daily values over the last 7 days of the 2-week run-in/wash-out (i.e., the last 7 days prior to the day of starting treatment period [Weeks 1-4/Weeks 7-10]).
Time Frame: Crossover Period Weeks 1-4, and 7-10
Population: PPS (Per Protocol Set): randomized subjects less those who did not complete treatment.
Measure: Mean (Standard Error); unit: Liters/minute
Groups:
- SFC 50/100 Mcg/Day: Per Protocol Set who received GW815SF (SFC, Salmeterol/Fluticasone propionate combination) HFA (Hydro Fluoro Alkane) MDI (Metered Dose Inhaler) 25/50 mcg twice daily
- SLM 50 Mcg + FP 100 Mcg/Day: Per Protocol Set who received SLM (Salmeterol) DPI (Dry Powder Inhaler) 25 mcg +FP (Fluticasone Propionate) DPI 50 mcg twice daily
Arm/Group | SFC 50/100 Mcg/Day | SLM 50 Mcg + FP 100 Mcg/Day
Number analyzed (Participants) | 48 | 48
Liters/minute | 14.3 (4.53) | 17.1 (4.53)
Statistical Analysis 1: Comparison: SFC 50/100 Mcg/Day vs SLM 50 Mcg + FP 100 Mcg/Day; Difference between treatments [(SLM + FP)- SFC](SE) 2.8 (5.91); Test type: Non-Inferiority or Equivalence — Equivalence margin + or - 15 L/min; p = 0.6383, Mixed Models Analysis — Confidence Interval; Mean Difference (Net) = 2.8, 95% CI [-9.10 to 14.69], Standard Error of Mean 5.91

2. Secondary Outcome: Adjusted Mean Change From Baseline in Percent Predicted Morning PEF(%) During the 4-week Treatment Periods
Description: Mean change from baseline = value at each assessment period (mean of the values obtained at each assessment period [Weeks 1-4/Weeks 7-10]) minus baseline value. Baseline: Mean of the daily values over the last 7 days of the 2-week run-in/wash-out.
Time Frame: Crossover Period Weeks 1-4, 7-10
Population: PPS
Measure: Mean (Standard Error); unit: Percentage of predicted value
Arm/Group | SFC 50/100 Mcg/Day | SLM 50 Mcg + FP 100 Mcg/Day
Number analyzed (Participants) | 48 | 48
Percentage of predicted value | 5.38 (1.543) | 6.73 (1.543)

3. Secondary Outcome: Adjusted Mean Change From Baseline in Percent Personal Best Morning PEF(%) During the 4-week Treatment Periods
Description: as for outcome 2
Time Frame: Crossover Period weeks 1-4, 7-10
Population: PPS
Measure: Mean (Standard Error); unit: Percentage of personal best value
Groups:
- SLM 50mcg + FP 100 Mcg/Day: Per Protocol Set who received SLM (Salmeterol) DPI (Dry Powder Inhaler) 25 mcg + FP (Fluticasone Propionate) DPI 50 mcg twice daily
Arm/Group | SFC 50/100 Mcg/Day | SLM 50mcg + FP 100 Mcg/Day
Number analyzed (Participants) | 48 | 48
Percentage of personal best value | 5.01 (1.480) | 6.46 (1.480)

4. Secondary Outcome: Adjusted Mean Change From Baseline in Evening PEF During the 4-week Treatment Periods
Description: as for outcome 2
Time Frame: Crossover Period weeks 1-4, 7-10
Population: PPS
Measure: Mean (Standard Error); unit: L/min
Arm/Group | SFC 50/100 Mcg/Day | SLM 50 Mcg + FP 100 Mcg/Day
Number analyzed (Participants) | 48 | 48
L/min | 16.3 (3.74) | 15.8 (3.74)

5. Secondary Outcome: Adjusted Mean Change From Baseline of Circadian Variation in Morning PEF(%) During the 4-week Treatment Periods
Description: as for outcome 2
Time Frame: Crossover Period Weeks 1-4, 7-10
Population: PPS
Measure: Mean (Standard Error); unit: Percentage of circadian variation
Arm/Group | SFC 50/100 Mcg/Day | SLM 50 Mcg + FP 100 Mcg/Day
Number analyzed (Participants) | 48 | 48
Percentage of circadian variation | 0.06 (0.638) | -0.08 (0.638)

6. Secondary Outcome: Percentage of Subjects With Symptom-Free Nights & Days
Description: Percentage of subjects with Symptom Free Nights & Days after 4 weeks of Treatment
Time Frame: Crossover Period Week 1-4, 7-10
Population: PPS
Measure: Number; unit: Percent of participants
Arm/Group | SFC 50/100 Mcg/Day | SLM 50 Mcg + FP 100 Mcg/Day
Number analyzed (Participants) | 48 | 48
Percent of participants
  Baseline | 72.9 | 81.3
  After 4 Weeks of Treatment | 91.7 | 81.3

7. Secondary Outcome: Percentage of Subjects With Rescue Medication-Free Nights and Days
Description: Percentage of subjects with Rescue Medication Free Nights & Days after 4 weeks of Treatment
Time Frame: Crossover Period Weeks 1-4, 7-10
Population: PPS
Measure: Number; unit: Percentage of participants
Arm/Group | SFC 50/100 Mcg/Day | SLM 50 Mcg + FP 100 Mcg/Day
Number analyzed (Participants) | 48 | 48
Percentage of participants
  Baseline | 87.5 | 87.5
  After 4 Weeks of Treatment | 93.8 | 87.5

8. Secondary Outcome: Adjusted Mean Change From Baseline in Morning PEF During the 20-week Extension Treatment Period
Description: Mean change from baseline = value at assessment period (mean of the values obtained at assessment period (Weeks 11-30).) minus baseline value. Baseline: Mean of the daily values over the last 7 days prior to the day of starting of the Extension period (Weeks 11-30).
Time Frame: Extension Period Weeks 11-30
Population: FAS (Full Analysis Set) during the Extension period: all subjects switched to Extension period and received GW815SF HFA MDI.
Measure: Mean (Standard Deviation); unit: L/min
Groups:
- SFC 50/100 Mcg/Day: Full Analysis Set who received GW815SF (SFC, Salmeterol/Fluticasone propionate combination) HFA (Hydro Fluoro Alkane) MDI (Metered Dose Inhaler) 25/50 mcg twice daily
Arm/Group | SFC 50/100 Mcg/Day
Number analyzed (Participants) | 50
L/min | 3.0 (24.56)

9. Secondary Outcome: Adjusted Mean Change From Baseline in Percent Predicted Morning PEF(%) During the 20-Week Extension Treatment Period
Description: Mean change from baseline = value at assessment period (mean of the values obtained at assessment period [Weeks 11-30]) minus baseline value. Baseline: Mean of the daily values over the last 7 days prior to the day of starting the Extension period (Weeks 11-30).
Time Frame: Extension Period weeks 11-30
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percentage of predicted value
Arm/Group | SFC 50/100 Mcg/Day
Number analyzed (Participants) | 50
Percentage of predicted value | 1.46 (9.568)

10. Secondary Outcome: Adjusted Mean Change From Baseline in Percent Personal Best Morning PEF(%) During the 20-week Extension Treatment Period
Description: as for outcome 9
Time Frame: Extension Period weeks 11-30
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percentage of personal best value
Arm/Group | SFC 50/100 Mcg/Day
Number analyzed (Participants) | 50
Percentage of personal best value | 1.29 (8.541)

11. Secondary Outcome: Adjusted Mean Change From Baseline in Evening PEF During the 20-week Extension Treatment Period
Description: as for outcome 9
Time Frame: Extension Period weeks 11-30
Population: FAS (Full Analysis Set) during the Exension period: all subjects switched to Extension period and received GW815SF HFA MDI.
Measure: Mean (Standard Deviation); unit: L/Min
Arm/Group | SFC 50/100 Mcg/Day
Number analyzed (Participants) | 50
L/Min | 2.7 (23.43)

12. Secondary Outcome: Adjusted Mean Change From Baseline of Circadian Variation in PEF(%) During the 20-Week Extension Treatment Period
Description: as for outcome 9
Time Frame: Extension Period weeks 11-30
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percentage of circadian variation
Arm/Group | SFC 50/100 Mcg/Day
Number analyzed (Participants) | 50
Percentage of circadian variation | -0.37 (3.568)

13. Secondary Outcome: Percentage of Subjects With Symptom-Free Nights & Days After 20 Weeks of Treatment
Description: Percentage of subjects with Symptom Free Nights & Days after 20 weeks of Treatment (at week 30).
Time Frame: Extension Period Weeks 11-30
Population: as for outcome 8
Measure: Number; unit: Percentage of participants
Arm/Group | SFC 50/100 Mcg/Day
Number analyzed (Participants) | 50
Percentage of participants
  Baseline | 84.0
  After 20 weeks of treatment (at week 30) | 84.8

14. Secondary Outcome: Percentage of Subjects With Rescue Medication-Free Nights & Days After 20 Weeks of Treatment
Description: Percentage of subjects with Rescue Medication Free Nights & Days after 20 weeks of Treatment (at week 30).
Time Frame: Extension Period Weeks 11-30
Population: as for outcome 8
Measure: Number; unit: Percentage of participants
Arm/Group | SFC 50/100 Mcg/Day
Number analyzed (Participants) | 50
Percentage of participants
  Baseline | 90.0
  After 20 weeks of treatment (at week 30) | 89.1

ADVERSE EVENTS:
Groups:
- SFC 50/100 Mcg/Day: Safety Population who received GW815SF (SFC, Salmeterol/Fluticasone Propionate combination) HFA (Hydro Fluoro Alkane) MDI (Metered Dose Inhaler) 25/50 mcg twice daily in Crossover Period Weeks 1-4 and 7-10
- SLM 50 + FP 100 Mcg/Day: Safety Population who received SLM (Salmeterol) DPI (Dry Powder Inhaler) 25 mcg +FP (Fluticasone Propionate) DPI 50 mcg twice daily in Crossover Period Weeks 1-4 and 7-10
- SFC 50/100mcg/Day (Extension Period): Safety Population who switched to Extension Period and received GW815SF HFA MDI 25/50mcg twice daily during the Extension period
Arm/Group | SFC 50/100 Mcg/Day | SLM 50 + FP 100 Mcg/Day | SFC 50/100mcg/Day (Extension Period)
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/50 | 0/51
Other Adverse Events (participants affected / at risk) | 12/51 | 10/50 | 35/51
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | SFC 50/100 Mcg/Day (N=51) | SLM 50 + FP 100 Mcg/Day (N=50) | SFC 50/100mcg/Day (Extension Period) (N=51)
Upper Respiratory Tract inflammation (Respiratory, thoracic and mediastinal disorders) | 7 | 3 | 17/50
Nasopharyngitis (Infections and infestations) | 2 | 4 | 7/50
Gastroenteritis (Infections and infestations) | 1 | 2 | 7/50
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 5/50
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 4/50
Stomatitis (Gastrointestinal disorders) | 2 | 0 | 3/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit an investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not preceed the primary publication of the entire clinical trial.